CLINICAL TRIAL: NCT02327026
Title: Initial Airway Management in Patients With Out-of-Hospital Cardiac Arrest: Tracheal Intubation vs. Bag-valve-mask Ventilation - CAAM STUDY
Brief Title: Tracheal Intubation vs. Bag-valve-mask Ventilation in Patients With Out-of-Hospital Cardiac Arrest _ CAAM STUDY
Acronym: CAAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130932; 2014-A01109-38 (Other: IDRCB)
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Out-of-hospital cardiac arrest; Bag-valve-mask ventilation; Tracheal intubation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bag-valve-mask ventilation (Experimental): Airway management including initial bag-valve-mask ventilation by the medical team during OHCA. When standard bag-valve-mask ventilation is possible, the patient will be intubated in case of a return of spontaneous circulation. When standard bag-valve-mask ventilation is impossible or in case of massive regurgitation of gastric content (after randomisation), intubation of patient is the preferred alternative
  Interventions: Procedure: bag-valve-mask ventilation
- tracheal intubation (Active Comparator): Tracheal intubation during OHCA by the medical team: The standard intubation procedure is to use a non-styletted tube and no sedation. When standard laryngoscopy-assisted intubation is not possible, an alternate procedure will be used based on the French consensus conference guidelines on difficult airway management.
  Interventions: Procedure: tracheal intubation

INTERVENTIONS:
Procedure: bag-valve-mask ventilation — Airway management including initial bag-valve-mask ventilation by the medical team during OHCA. When standard bag-valve-mask ventilation is possible, the patient will be intubated in case of a return of spontaneous circulation. When standard bag-valve-mask ventilation is impossible or in case of massive regurgitation of gastric content (after randomisation), intubation of patient is the preferred alternative.
  Arms: bag-valve-mask ventilation
Procedure: tracheal intubation — Tracheal intubation during OHCA by the medical team: The standard intubation procedure is to use a non-styletted tube and no sedation. When standard laryngoscopy-assisted intubation is not possible, an alternate procedure will be used based on the French consensus conference guidelines on difficult airway management
  Arms: tracheal intubation

SUMMARY:
The aim of this study is to improve the management of patients in cardiac arrest, and this by comparing two initial airway management methods: Tracheal intubation and bag-valve-mask ventilation.

The survival rate at 28-day with favorable neurological function will be compared in the tracheal intubation group versus the bag-valve-mask group

DETAILED DESCRIPTION:
It is a multicenter prospective non-inferiority open randomized controlled trial in patients with out-of-hospital cardiac arrest carried out in physician-staffed emergency medical services.

The investigators hypothesis is that basic airway management (i.e. bag-valve-mask ventilation) is safe and may avoid the deleterious effects of tracheal intubation including interruption of chest compressions.

On medical team's arrival at the scene and after verification of participant's eligibility, patients will be enrolled in the study and randomly assigned to either initial bag-valve-mask ventilation or tracheal intubation. After the hospital admission, all patients will be intubated whatever the initial airway management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Patient with out-of-hospital cardiac arrest on medical team's arrival
* Resuscitation attempted
* Medical insurance

Exclusion Criteria:

* Massive suspected aspiration
* Presence of do-not-resuscitate order
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2043 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Survival with favorable neurological function defined as Glasgow-Pittsburgh Cerebral Performance Categories (CPC) of 2 or less. | Day 28
  Survival at 28-day with favorable neurological function defined as Glasgow-Pittsburgh Cerebral Performance Categories (CPC) of 2 or less. In case of neurological disability before randomization, the survival associated the same degree of disability will be considered a favorable neurological function

SECONDARY OUTCOMES:
Survival at hospital admission | Day 0
Survival | Day 28
Survival at hospital discharge | up to Day 28
Neurologic outcomes assessed by modified Rankin scale score | Day 28
Rate of return of spontaneous circulation (ROSC) | Day 0
Intubation difficulty assessed by Intubation difficulty Scale score | Day 0
Complications related to tracheal intubation | Day 0
  Complications related to tracheal intubation during advanced Cardiopulmonary Resuscitation (CPR): failure, esophageal intubation, mainstem intubation, vomiting, pulmonary aspiration, dental trauma, extubation
Complications related to bag-valve-mask ventilation | Day 0
  Complications related to bag-valve-mask ventilation during advanced CPR: regurgitation of gastric content
Technique's failure defined as mortality | Day 0, Day 28
  Technique's failure defined as mortality at 28-day or regurgitation during the procedure or failure of the procedure (failure to ventilate in the bag-valve-mask ventilation or failure to intubate in the intubation group)
Ventilation difficulty with bag-valve-mask measured with a visual-analog-scale (VAS) | Day 0
Han's mask ventilation classification | Day 0
Difficult mask ventilation signs | Day 0
Time to completion of tracheal intubation (TI) procedure | Day 0
  Time to completion of tracheal intubation (TI) procedure measured from the instant that the laryngoscope blade touches the patient to the moment that the tracheal tube cuff is inflated
Duration of the interruption of chest compression during TI procedure | Day 0
  Duration of the interruption of chest compression during TI procedure
Duration of the interruption of chest compression during advanced CPR (from medical team's arrival to decision to stop CPR) | Day 0
  Duration of the interruption of chest compression during advanced CPR (from medical team's arrival to decision to stop CPR)
Duration of advanced CPR | Day 0
  Duration of advanced CPR (from medical team's arrival to decision to stop CPR)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ADNET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Avicenne Hospital - Aphp, Bobigny, Île-de-France Region, France

REFERENCES:
- [Derived] Jabre P, Penaloza A, Pinero D, Duchateau FX, Borron SW, Javaudin F, Richard O, de Longueville D, Bouilleau G, Devaud ML, Heidet M, Lejeune C, Fauroux S, Greingor JL, Manara A, Hubert JC, Guihard B, Vermylen O, Lievens P, Auffret Y, Maisondieu C, Huet S, Claessens B, Lapostolle F, Javaud N, Reuter PG, Baker E, Vicaut E, Adnet F. Effect of Bag-Mask Ventilation vs Endotracheal Intubation During Cardiopulmonary Resuscitation on Neurological Outcome After Out-of-Hospital Cardiorespiratory Arrest: A Randomized Clinical Trial. JAMA. 2018 Feb 27;319(8):779-787. doi: 10.1001/jama.2018.0156. PMID 29486039